CLINICAL TRIAL: NCT06090929
Title: STN-DBS is a Risk Factor of Sialorrhea in Patients With Advanced Parkinson's Disease
Brief Title: STN-DBS and the Risk of Sialorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: DBS & drooling in PD
Record Dates: First submitted 2023-10-07; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Deep Brain Stimulation; Sialorrhea
MeSH Terms: conditions — Parkinson Disease; Sialorrhea

STUDY DESIGN:
Intervention Model Description: A total of 234 participants were enrolled between June 2019 and July 2021; 198 patients with PD receive STN-DBS (n=99) or medication (n=99)
Who Masked: Investigator
Masking Description: Investigator was blinded to the status of DBS or non-DBS during the scoring of DRS, DSFS and drooling rate examination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with STN-DBS (Experimental): Patients accepted DBS implanted at the baseline
  Interventions: Device: STN-DBS
- Patients without STN-DBS (No Intervention): Patients only accepted medication treatment before the end point

INTERVENTIONS:
Device: STN-DBS — STN-DBS was implanted according normal process
  Arms: Patients with STN-DBS

SUMMARY:
OBJECTIVE: The aims of this study were to assess the incidence rate and risk factors for sialorrhea in the long-term follow-up in a cohort of 170 patients with advanced Parkinson's disease [84 with deep brain stimulation (DBS) and 86 on medical treatment].

Design, setting, and participants: This study was a multi-center prospective non-randomized concurrent clinical trial. A total of198 persons with Parkinson disease were referred for DBS between June 2019 and July 2021 and analyzed between June 2023 and July 2023.The primary outcome follow-up visit was conducted 36 months after DBS.

DETAILED DESCRIPTION:
IMPORTANCE: Sialorrhea is a frequent and disabling symptom in patients with PD. No prospective study has been specifically designed to test the effects of DBS on sialorrhea development.

OBJECTIVE: The aims of this study were to assess the incidence rate and risk factors for sialorrhea in the long-term follow-up in a cohort of 170 patients with advanced Parkinson's disease [84 with deep brain stimulation (DBS) and 86 on medical treatment].

Design, setting, and participants: This study was a multi-center prospective non-randomized concurrent clinical trial. A total of198 persons with Parkinson disease were referred for DBS between June 2019 and July 2021 and analyzed between June 2023 and July 2023.The primary outcome follow-up visit was conducted 36 months after DBS.

INTERVENTIONS: Bilateral subthalamic nucleus DBS was performed in one study arm and not performed in the other. Both arms of the study completed the drooling rating scale (DRS), the drooling severity and frequency scale (DSFS) and examination of salivary secretion rate.

MAIN OUTCOMES AND MEASURES: The primary outcome was the DRS scores of the patients with PD, with or without STN-DBS 36 months postoperatively. The secondary outcomes included the DSFS scores, saliva secreting rate, ratio of botox injection in different group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Age between 20 and 80 years
* without drooling
* swallowing function <5 on the Drooling Rate Scale (DRS).
* Medications affecting drooling had to have stopped medications at least 4 weeks before study entry.

Exclusion Criteria:

* Not he typical PD
* Subjects on warfarin,
* with significant medical illnesses or neuromuscular transmission disorders
* past use of BoNT
* -cognitive impairment (<23/30 on Mini Mental Status Exam) were excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
DRS score 36 months postoperatively | 36 months after STN-DBS
  Drooling Rate Scale (DRS) which range from 0 to 15 was used to evaluate the status of drooling. 0 stands for non-drooling and 15 stands for the severe status of drooling

SECONDARY OUTCOMES:
DSFS score 36 months postoperatively | 36 months after STN-DBS
  drooling severity scale (DSFS) which range from 0 to 5 was used to evaluate the status of drooling. 0 stands for non-drooling and 5 stands for the severe status of drooling
BOTOX injection ratio 36 months postoperatively | 36 months after STN-DBS or a longer follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Chao Zhang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data (IPD) could be available to other researchers on request without business benefits.

REFERENCES:
- [Derived] Sun J, Cheng L, Li Z, Jia J, Wu Q, Hou Y, Wang Q, Zhang G, Wang H, Li X, Li W, Zhang C. Deep brain stimulation of the subthalamic nucleus increases the risk of sialorrhea in patients with advanced Parkinson's disease. Parkinsonism Relat Disord. 2024 Jun;123:106075. doi: 10.1016/j.parkreldis.2024.106075. Epub 2024 Mar 9. PMID 38492517